CLINICAL TRIAL: NCT06407583
Title: ProMIO 2.0; A Powerful Lifestyle Intervention for Older Adults From Ethnic Minorities
Brief Title: ProMIO2.0; A Powerful Lifestyle Intervention for Older Adults From Ethnic Minorities
Acronym: ProMIO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ProMIO2.0 - NL75885.029.21; RAAK.MKB12.033 (Other Grant/Funding Number: NWO - SIA Raak)
Record Dates: First submitted 2023-07-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenia; Diabetes; Overweight; Ethnic Minorities; Musculoskeletal Diseases
Keywords: Lifestyle intervention; Protein; Multicomponent exercise; Older adults; Ethnic minorities
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus; Overweight; Musculoskeletal Diseases

STUDY DESIGN:
Intervention Model Description: The design is a single blind parallel RCT with a control group and intervention group. The study duration is 6 months.
  Control: no intervention (education only) Intervention: ProMIO2.0 lifestyle program including multicomponent exercise and protein intake counselling.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Participants receiving regular care in the 6 months period. They receive a brief education session at start about exercise and protein.
- ProMIO2.0 intervention group (Experimental): Participants receiving regular care and our newly developed lifestyle intervention for 6 months period. The intervention is culture specific and contains of:
  * Dietetic care focused on protein intake (protein counselling)
  * Multicomponent exercise (physical therapy); a combination between group sessions and home-based exercise
  The first 3 months are intensive phase, second 3 months guidance gradually decreases.
  Interventions: Behavioral: ProMIO2.0 program

INTERVENTIONS:
Behavioral: ProMIO2.0 program — ProMIO2.0 is a lifestyle intervention carried out by physiotherapy and dietetics. They guide and encourage the participants to achieve the following behavioral goals:
  * moderate/intensive exercise (e.g. walking) for 150-300 minutes per week
  * Muscle-strengthening exercises 2x a week
  * Supplemented with balance and flexibility exercises
  * 1.2 grams of protein per kilogram of body weight per day (~25-30 grams of protein per meal, 4x/day) The combination of consultations, information sessions and on-site training at the physiotherapist should ensure that participants acquire the necessary knowledge, awareness and skills to adopt the health behavior in daily life. Materials such as posters, pedometers and videos are used for support.
  The intervention is divided into 2 phases, which indicate the degree of professional guidance:
  1. intensive guidance (month 0 - 3)
  2. average guidance (months 4 - 6)
  Arms: ProMIO2.0 intervention group

SUMMARY:
Older adults from ethnic minorities show on average a worse disease risk profile compared to the majority populations. An important risk factor to develop chronic diseases is the loss of muscle mass and functioning, also known as sarcopenia. Several randomized controlled trials (RCTs) showed that the combination of adequate protein intake and physical exercise is most effective to prevent the loss of muscle mass, strength and functioning in older adults. However, until shortly, no intervention that included protein and exercise was available that accounted for the special socio-cultural needs of ethnic minority populations. Therefore the Amsterdam University of Applied Sciences (AUAS) and ProMIO project group developed a cultural sensitive lifestyle intervention with protein and exercise carried out by dieticians and physical therapists to provide a tailored treatment for older adults from ethnic minorities. This project aims to evaluate the effectiveness of this new intervention on protein intake, physical activity behavior, muscle mass, muscle strength, function and quality of life. The cost-effectiveness of this new intervention will also be evaluated.

DETAILED DESCRIPTION:
Primary Objective: To investigate the effectiveness of the ProMIO lifestyle intervention (targeting protein intake and exercise behavior) on physical functioning, in older adults from ethnic minorities (Surinamese).

The intervention will be a lifestyle intervention targeted at changing health behaviors in older adults from ethnic minorities in the Netherlands. Methods will be used that target specific behavioral determinants in order to optimize both exercise and dietary behavior. We aim to reach the following behavioral outcomes:

* 1.2g/kg BW/day (~25 - 30 grams of protein per meal (4x/day))
* Reaching the WHO physical activity guidelines for older adults:

  * At least 150-300 minutes/week moderate-intensity aerobic physical activity (such as walking)
  * 2x/week strength, balance and functional exercises

Based on previous research it is expected that by optimizing these health behaviors, muscle mass, muscle strength, and physical functioning will improve.

Secondary Objective(s):

* To investigate the effectiveness of the ProMIO lifestyle intervention (targeting protein intake and exercise behavior) on muscle mass and muscle strength, in older adults from ethnic minorities
* To investigate the effectiveness of the ProMIO lifestyle intervention on protein intake and physical activity behavior in older adults from ethnic minorities
* To investigate the cost-effectiveness of the ProMIO lifestyle intervention in comparison to an health education intervention.

The (cost-)effectiveness of the ProMIO intervention will be investigated using a single blind randomized controlled trial (RCT) with two parallel arms.

First, potential participants will be recruited and screened for eligibility. Secondly, participants will be randomly assigned to one of the two groups; the intervention group or the control group.

The full study will comprise a 6-month intervention, divided in two phases, and consisting of a multicomponent exercise training (MCE) program provided by physical therapists and a protein intervention provided by dieticians. Each participant will be supervised and monitored by a physical therapist and a dietician, who are providing regular consulting sessions.

Exercise activities, like group exercise training, will be provided by certified trainers and health education will be provided by AUAS graduate students with a background in nutrition and/or physical exercise. Certified trainers and graduate students are supervised and guided by the physical therapist and dietician. The intensity of the professional support during the intervention will be highest in the first phase and taper off during the second phase. Participants are expected to adopt most of the desired behavioral activities in daily living without professional help. Data will be collected at baseline (T1) and after 3 (T2), and 6 (T3) months.

Outcome measures are a combination between quantitative and qualitative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Born in Surinam (or at least one of the parents was born there)
* Aged ≥55 years
* Physical ability and willingness to execute an MCE program
* Ability and willingness to comply with the study protocol
* Written informed consent
* Consent of the study physician

Exclusion Criteria:

* Aged <55 years
* Diagnosed with renal insufficiency (MDRD<30, GP approved)
* Suffering from physical disabilities causing the inability to perform the main exercises (walking aids or mild visual impairment are not an exclusion criteria)
* Diagnosed unstable coronary heart disease (CHD), decompensated heart failure, or uncontrolled arrhythmias
* End stage Chronic Obstructive Pulmonary Disease (COPD) GOLD >3
* Phase IV cancer
* Diagnosed degenerative neurocognitive disorders
* Active (para-)medical treatment interfering with this intervention
* Current enrolment in a fixed rehabilitation program or other intervention studies
* Palliative treatment or a life expectancy of ≤3 months
* A trip >2 weeks planned in first three months of study or >2 months during the rest of the intervention period

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 76 (Actual)
Dates: Start 2022-05-24 (Actual); Primary Completion 2023-06-08 (Actual); Study Completion 2023-06-08 (Actual)

PRIMARY OUTCOMES:
Physical functioning | baseline, 3 months
  change in meters from baseline to 3 months by 6 Minute Walk Test
Physical functioning | baseline, 6 months
  change in meters from baseline to 6 months by 6 Minute Walk Test

SECONDARY OUTCOMES:
30-sec Chair Stand Test | baseline, 3 months, 6 months
  (frequency) change from baseline to 3 or 6 months
Balance (Single Leg Stand Test) | baseline, 3 months, 6 months
  (seconds) - change from baseline to 3 or 6 months
Strenght (1RM with Microfet) | baseline, 3 months, 6 months
  (kg) change from baseline to 3 or 6 months
Strenght with Hand Grip Strenght | baseline, 3 months, 6 months
  (kg) change from baseline to 3 or 6 months
Body composition Lenght | baseline, 3 months, 6 months
  (meters) change from baseline to 3 or 6 months
Body composition Weight | baseline, 3 months, 6 months
  (kg) change from baseline to 3 or 6 months
Body composition BMI | baseline, 3 months, 6 months
  (kg/m2) change from baseline to 3 or 6 months
Body composition 2D muscle echo | baseline, 3 months, 6 months
  (cm2) change from baseline to 3 or 6 months
Behavioral outcome - Dietary intake (48h recall) | baseline, 3 months, 6 months
  macronutrient and micronutrient change from baseline to 3 or 6 months
Behavioral outcome - Physical Activity | baseline, 3 months, 6 months
  (PAMscore) - change from baseline to 3 or 6 months
Quality of Life (QoL) | baseline, 3 months, 6 months
  (score) change from baseline to 3 or 6 months
Sarcopenia screening (SarQoL) | baseline, 3 months, 6 months
  (score) change from baseline to 3 or 6 months
Frailty | baseline, 3 months, 6 months
  (score) change from baseline to 3 or 6 months
Activities of Daily Living (ADL) Katz | baseline, 3 months, 6 months
  (score) change from baseline to 3 or 6 months
Pain (NRS) | baseline, 3 months, 6 months
  (NRS) change from baseline to 3 or 6 months
Sleep (NRS) | baseline, 3 months, 6 months
  (NRS) change from baseline to 3 or 6 months
Risk of Falls (NRS) | baseline, 3 months, 6 months
  (NRS) change from baseline to 3 or 6 months
Efficacy Scale International (sFES-I) | baseline, 3 months, 6 months
  (score) change from baseline to 3 or 6 months
symptoms of depression (CES-D) | baseline, 3 months, 6 months
  (score) change from baseline to 3 or 6 months
Cost effectiveness - Productivity Cost Questionnaire (PCQ) | baseline, 6 months
  (score) change from baseline to 6 months
Cost effectiveness - Cost of Quality (MCQ) | baseline, 6 months
  (score) change from baseline to 6 months
Process evaluation | 6 months
  Process evaluation questionnaire and focus group sessions
Social democrafic characteristics | screening, baseline
  e.g. age (years), gender (f/m), highest education level
Medical history | screening
  all medical events and diseases reported
Medication use | screening and during study
  all medication reported at start and during the trial
Adverse events | During study
  all adverse events reported during the intervention study
Adherence to the intervention | During study
  Specified for exercise routine and protein intake; a % of attendance and minimal 1.2 g/kgBW/day protein intake

CONTACTS AND LOCATIONS:
Overall Officials: Peter Weijs, Prof Dr Ir, Principal Investigator — Amsterdam University of Applied Sciences
Locations (1):
- Amsterdam University of Applied Sciences, Center of Expertise Urban Vitality, Amsterdam, N-H, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Restricted on Figshare following our OpenScience regulations
Supporting Information: Study Protocol, ICF, CSR
Time Frame: After study completion
Access Criteria: Restricted untill publication.

REFERENCES:
- [Derived] Biersteker EJM, van den Helder J, van der Spek N, Holwerda M, Kruizenga H, Weijs PJM, Tieland M. Culture-sensitive lifestyle intervention tailored to non-Western migrant older adults improves physical performance: A randomized controlled trial. J Nutr Health Aging. 2025 Aug;29(8):100584. doi: 10.1016/j.jnha.2025.100584. Epub 2025 May 22. PMID 40409139
- See also: Webpage of our institute — https://www.hva.nl/urban-vitality/gedeelde-content/projecten/voeding-en-beweging/promio-2.0.html
- See also: Webpage of our nutrition and exercise platform — https://voedingenbeweging.nu/project/promio/